CLINICAL TRIAL: NCT04490551
Title: Combining Risk Factors and Faecal Immunochemical Testing in Colorectal Cancer Screening: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AMC_MDL_161
Record Dates: First submitted 2020-07-13; First posted 2020-07-29 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Neoplasms; Colorectal Adenoma; Colorectal Adenoma and Carcinoma
Keywords: Colorectal Cancer; Screening; Model; Faecal Immunochemic Test; FIT; Occult Blood; Risk Factors; Logistic Regression; Advanced Neoplasia; Advanced Adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma

STUDY DESIGN:
Intervention Model Description: The researchers conduct a parallel group randomized controlled trial. Asymptomatic individuals will be randomized to either risk-based screening or FIT-only screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will be screened with the risk-based model. The input of the model will be gathered with the FIT, a validated questionnaire, and from data of the Dutch general population registry. The threshold of the model will be set at a calculated risk of 0.10. To comply with ethical guidelines, all participants in this group with a FIT result of >=15 mcg Hb/g faeces and a calculated risk of <0.10 will also be offered a colonoscopy.
  Interventions: Diagnostic Test: Risk-based logistic regression model; Diagnostic Test: FIT
- Control group (Active Comparator): This group will be screened with the FIT. The threshold of the FIT will be set at >= 15 mcg Hb/g faeces.
  Interventions: Diagnostic Test: FIT

INTERVENTIONS:
Diagnostic Test: Risk-based logistic regression model — The intervention will be a risk-based logistic regression model that takes multiple variables into account to calculate the risk of advanced neoplasia as an outcome.
  Arms: Intervention group
Diagnostic Test: FIT — FIT is a stool-based test that detects human blood in faeces.
  Other Names: Faecal Immunochemic Test

SUMMARY:
Colorectal Carcinoma (CRC) is the third most frequent diagnosed cancer worldwide, with 1.4 million new cases every year. In an attempt to reduce this number many countries have implemented a nationwide screening programme targeted at detecting CRC in an early phase using fecal immunochemical tests (FITs). People with an elevated level of blood in their stool are offered a colonoscopy, an invasive medical procedure where CRCs and premalignant lesions (together also referred to as advanced neoplasia) can be detected accurately.

However, the current screening method using FIT is not optimal. In FIT-based CRC screening studies, 1 in 4 participants with CRC and 2 in 3 participants with advanced neoplasia receive a negative FIT result. In contrast, an estimated 1 in 2 FIT-positives have advanced neoplasia at colonoscopy.

Recent studies have demonstrated that a risk model that takes into account the FIT result and other risk factors for CRC could enhance the effectiveness of a FIT-based CRC screening programme.

The objective of this study is to assess the yield of advanced neoplasia in the colon and rectum of a FIT-based risk model at colonoscopy, compared to that of a FIT-only CRC screening strategy. Our hypothesis is that a risk-based model yields significantly more advanced neoplasia at colonoscopy than the FIT by itself, and that it does not affect participation rate.

To assess this hypothesis, the investigators have designed a clinical trial in which the investigators randomize 23,000 asymptomatic individuals between the age of 55 and 75 years old to either risk-based screening (intervention group) or FIT-only screening (control group). The intervention group will receive a questionnaire on risk factors of CRC (e.g. smoking, family history of CRC), and a FIT. The control group will only receive the FIT. The positivity threshold of the FIT in both groups will be set at 15 micrograms haemoglobin per gram faeces. The positivity threshold of the risk-based model in the intervention group will be set at 0.10 (out of a range of 0 to 1), a threshold that is calculated with a goal to match the positivity rate of the control group.

Participants with a result that is above the thresholds of the FIT and/or the risk-based model will be invited to undergo a colonoscopy according protocol of the Dutch national screening program. After the study has ended, the investigators will compare both groups to assess our hypotheses.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Colorectal Cancer (CRC) is the third most frequent diagnosed cancer worldwide, with 1.4 million new cases every year. Mortality of CRC is estimated at around 40%. To reduce the incidence of CRC and to abate the negative consequences associated with CRC, methods for early detection of (pre)malignant colorectal lesions have extensively been researched and implemented. Colonoscopy is the reference standard for the detection of advanced neoplasia, but it requires trained endoscopists, carries a high burden, harbours a risk for complications in patients, and increases societal costs.

Most screening programs use methods to select screening participants with a high risk of advanced neoplasia for colonoscopy. One such method is the detection of blood in stool with faecal immunochemical tests (FITs).

Multiple nation-wide screening programs have now been implemented using FIT, including one in the Netherlands. In the Dutch CRC screening program, using a FIT threshold of 47 µg Hb/g faeces, the sensitivity of FIT in detecting CRC is 85.5%. The sensitivity of FIT in detecting advanced neoplasia (AN) is however substantially lower: 38%.

FIT-based screening also generates a high number of false positives, leading to unnecessary colonoscopies and distress for those patients. Approximately 1 in 2 FIT-positives has advanced neoplasia; the first round of the Dutch CRC screening program, using a FIT threshold of 47 µg Hb/g faeces, reached a positive predictive value of 54%.

Previous studies have demonstrated the existence of clinical risk factors for CRC, such as male gender, age, family history of CRC, and smoking. In a ZonMW sponsored project (ZonMW 50-50115-96-521) our group has shown that higher age, male sex, a family history with close relatives in whom CRC was diagnosed, and active smoking were all associated with the presence of advanced neoplasia (Stegeman et al, Gut, 2014).

Multiple CRC risk models have been developed using these risk factors, but most show only weak discriminatory power. Others have proposed risk models that additionally included molecular markers, increasing performance and discriminatory power, but these markers can be cumbersome to collect and can be costly in respect to the relative cheap FIT test. the investigators propose to combine CRC risk factors with the quantitative FIT result. FIT is a quantitative test with a variable cut-off level, and individuals with higher values of faecal haemoglobin are at higher risk of having advanced neoplasia at the cost of a lower specificity. Therefore, the quantitative result can be used as a weight-factor in a risk model.

Based on information on these risk factors for CRC and the quantitative FIT-result, our FIT-based risk model for CRC screening calculates the personal risk of having advanced neoplasia at colonoscopy. Inviting screening participants with elevated risk for colonoscopy, rather than those whose FIT result exceeds a pre-specified threshold, has the potential to increase the effectiveness and efficiency of FIT-based CRC screening. However, this requires participants to complete the questions about risk.

Our hypothesis is that integration of FIT score with known risk factors (age, gender, smoking, and family history of CRC) improves the number of participants in whom advanced neoplasia is detected, relative to the number of invitees. The investigators will compare a risk-based approach to screening, as described above, to the conventional FIT-only screening in a randomized controlled screening trial.

OBJECTIVES The study hypothesis is that risk-based CRC screening significantly outperforms FIT-only CRC screening in terms of the relative number of invitees in whom advanced neoplasia is detected at colonoscopy.

Primary Research Question: does risk-based CRC screening result in a higher relative number of invitees in whom advanced neoplasia is detected at colonoscopy compared to FIT-only CRC screening?

Secondary Research Questions:

i) Does risk-based CRC screening result in a higher standardized screening yield in whom advanced neoplasia is detected at colonoscopy compared to FIT-only CRC screening? ii) Is the participation rate of risk-based CRC screening non-inferior compared to FIT-only screening? iii) Does risk-based CRC screening result in a higher relative number of invitees in whom advanced neoplasia is detected at colonoscopy compared to FIT-only CRC screening at higher FIT-positivity thresholds (from 15 µg Hb /g faeces)? iv) Does risk-based CRC screening result in a higher relative number of invitees in whom proximally located advanced neoplasia is detected at colonoscopy compared to FIT-only CRC screening?

METHODS The investigators will perform a randomized controlled trial in 23,000 randomly selected men and women (aged 55 to 75 years) eligible for participation in the national CRC screening programme. All eligible participants will be second time invitees, living within a 25 km radius from the colonoscopy centre Bergman Clinics Amsterdam, which is accredited for the national population screening program.

Eligible individuals are randomly allocated on a 1:1 basis to an invitation for either risk-based CRC screening (intervention group) or FIT-only screening (control group). Randomization per household will be done before invitation. Study invitations are sent out by Foundation of Population Screening Mid-West (BoMW) early November 2019 before sending the FIT sample kit of the national screening program to the study cohort from January 2020 to April 2020. The study invitation is combined with a leaflet containing information on study participation. It will also contain an informed consent form, and a one-page questionnaire (if allocated to the intervention arm) with a self-addressed envelope to the research facility. The informed consent form will bear a unique study identification code.

The model that the investigators will use in this study for risk-based screening is derived from a model developed in a primary colonoscopy screening trial (Stegeman et al, Gut, 2014). The investigators have re-evaluated our multivariable risk model for CRC, with the aim to simplify it for daily practice. A number of risk factors (such as elements from diet) added little to the performance of the model, whereas collecting the necessary information proved rather tedious. The quantitative FIT result, age, sex, family history and smoking behaviour were the most decisive factors in the model.

This simplified FIT-based risk model had a performance like that of the extended model in the development dataset. In this study the investigators will calculate the risk of harbouring advanced neoplasia with our simplified FIT-based risk model, based on the quantitative FIT result, age, sex, family history and smoking behaviour (see below). The threshold and expected positivity rate of the risk-based model will be matched to the expected positivity rate of the FIT-only group.

Regression equation of the updated model:

ln(odds AN) = -4.955073942+0.9196052173*Smoking+0.3364761549* √FIT+0.370575346*family history of CRC-0.006934851*FIT+0.0228752117*age+0.070972656*gender

Probability of advanced neoplasia:

P (AN)=e^((odds AN))/(1+e^((odds AN))) If invitees that are allocated to the intervention group (i.e. questionnaire and FIT) only return the questionnaire, they do not qualify for a colonoscopy. When consenting invitees in the intervention group prefer not to complete the questionnaire, FIT tests will be analysed at a cut-off of 15 µg Hb/g faeces.

The type of FIT that will be used is the one used in the Dutch national screening programme: FOB-Gold (Sentinel, Italy). FIT-analyses and sending of FIT results will be performed according to the logistics as being used in the national screening. The FIT result and the result of the questionnaire will be entered in a database, to calculate the participant's risk. All FIT positives (≥15 µg Hb/g faeces) will be referred for consultation for colonoscopy at regional endoscopic centres. For the purpose of this study, FIT-negative but risk-positive participants (i.e. the combination of the results of the questionnaire and the quantitative FIT result) will also be invited for consultation for colonoscopy.

Colonoscopy will be performed by endoscopists accredited for our national screening programme and according to national and international quality guidelines. Quality indicators and endoscopic findings will be systematically recorded in a database, according to the standards of the national screening programme. Lesions will be immediately removed, if possible, and otherwise biopsies will be obtained. Histopathological assessment of these tissue samples will provide a definitive diagnosis. Data on location, size, macroscopic aspect, morphology and polypectomy will be recorded for all colonic lesions, which will be collected and evaluated by an accredited GI-pathologist according to the Vienna criteria. Advanced adenomas are defined as adenomas larger than 10 mm, adenomas with high-grade dysplasia or adenomas with a villous component of at least 25%. Advice regarding surveillance colonoscopy after removal of adenomatous polyps, large (≥10 mm) serrated lesions or cancer will be given to the clients according to the Dutch CBO consensus.

Screening invitees can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a screening invitee from the study for urgent medical reasons.

STATISTICAL ANALYSIS

Primary outcome The difference in screening yield will be estimated and expressed as an absolute difference per 1,000 invitees, with 95% confidence intervals. The investigators will test the null hypothesis of no difference in yield between the intervention and control group using the chi-square test.

Secondary outcome The standardized screening yield will be calculated by ranking participants according to their calculated risk (in risk-based screening) and comparing the yield of risk-based screening for the number of positives that matches the number of FIT-positives with FIT-only screening with a chi-square test. Additionally, the investigators will use the McNemar test statistic to test the null hypothesis of no gain in screening yield in the intervention group only, where the investigators can compare referrals based on FIT only with referrals based on FIT and calculated risk.

The participation rate will be calculated through the number of participants relative to the number of invitees in each arm. Differences in participation rate will be assessed using the chi square test. The difference in screening yield of proximally located advanced neoplasia between both arms will be estimated and expressed as an absolute difference per 1,000 invitees (with 95% confidence intervals). The null hypothesis of no difference in yield will be tested using the chi square test.

Statistical significance level P-values of lower than 0.05 will be considered statistically significant. All analysis between both arms are based on the intention-to-screen principle, unless stated otherwise. Statistical analyses will be performed using R.

Additional outcomes Model performance in comparison to the FIT will be assessed with the net reclassification improvement (NRI). In addition, the yield of the FIT-based risk model and the FIT will be assessed at a broad range of FIT thresholds and will be estimated and expressed as the number of detected advanced neoplasia per 1,000 invitees (intention-to-screen) and per 1,000 colonoscopies (per protocol). Differences in the yield will be tested using a chi square test. Any missing data that was intended to be used as input for the risk-model, will be classified as '0'.

ETHICAL CONSIDERATIONS The study will be conducted according to the principles of the Declaration of Helsinki (Version October 2008) and the Population Screening Act (WBO). Permission to conduct this study has been granted by the Dutch Health Council and the Dutch Minister of Healthcare.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a screening invitee must meet the following criteria:

1. The screening invitee must be at least 55 years old, and no older than 75 years old, at the day of invitation by the Foundation of Population Screening Mid-West
2. The screening invitee must be eligible for participation in the second round of the Dutch CRC Population Screening Programme
3. The screening invitee must return a signed informed consent form

Exclusion Criteria:

A potential screening invitee who meets any of the following criteria will be excluded from participation in this study:

1. if he or she receives active treatment for CRC and/or AN, including palliative care.
2. if he or she fails to return a sample that is adequate for FIT testing.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Females
Enrollment: 6753 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Yield of Advanced Neoplasia | 10 weeks
  The primary outcome is the yield of advanced neoplasia, defined as the relative number of invitees in whom advanced neoplasia is detected at colonoscopy.

SECONDARY OUTCOMES:
Standardized Screening Yield | 10 weeks
  standardized screening yield: ranking the number of participants according to their calculated risk and comparing the yield of risk-based screening for the number of positives that matches the number of FIT-positives with FIT-only screening.
Participation Rate | 10 weeks
  participation rate, defined as the relative number of invitees participating in screening.
Yield of Advanced Neoplasia at Other Thresholds | 10 weeks
  yield of advanced neoplasia, defined as the relative number of invitees with advanced neoplasia detected at colonoscopy, at FIT-positivity thresholds of 15 µg Hb/g faeces and higher.
Yield of Proximally Located Advanced Neoplasia | 10 weeks
  yield of proximally located advanced neoplasia, defined as the relative number of referred participants in whom proximally located advanced neoplasia is detected at colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, PhD MD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, locatie Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Conditional on the permission of the Dutch government, anonymized research data may be shared after publication of the results in a peer-reviewed paper.

REFERENCES:
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Winawer S, Fletcher R, Rex D, Bond J, Burt R, Ferrucci J, Ganiats T, Levin T, Woolf S, Johnson D, Kirk L, Litin S, Simmang C; Gastrointestinal Consortium Panel. Colorectal cancer screening and surveillance: clinical guidelines and rationale-Update based on new evidence. Gastroenterology. 2003 Feb;124(2):544-60. doi: 10.1053/gast.2003.50044. PMID 12557158
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Kronborg O, Fenger C, Olsen J, Jorgensen OD, Sondergaard O. Randomised study of screening for colorectal cancer with faecal-occult-blood test. Lancet. 1996 Nov 30;348(9040):1467-71. doi: 10.1016/S0140-6736(96)03430-7. PMID 8942774
- [Background] Hewitson P, Glasziou P, Watson E, Towler B, Irwig L. Cochrane systematic review of colorectal cancer screening using the fecal occult blood test (hemoccult): an update. Am J Gastroenterol. 2008 Jun;103(6):1541-9. doi: 10.1111/j.1572-0241.2008.01875.x. Epub 2008 May 13. PMID 18479499
- [Background] Hewitson P, Glasziou P, Irwig L, Towler B, Watson E. Screening for colorectal cancer using the faecal occult blood test, Hemoccult. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD001216. doi: 10.1002/14651858.CD001216.pub2. PMID 17253456
- [Background] Allison JE, Sakoda LC, Levin TR, Tucker JP, Tekawa IS, Cuff T, Pauly MP, Shlager L, Palitz AM, Zhao WK, Schwartz JS, Ransohoff DF, Selby JV. Screening for colorectal neoplasms with new fecal occult blood tests: update on performance characteristics. J Natl Cancer Inst. 2007 Oct 3;99(19):1462-70. doi: 10.1093/jnci/djm150. Epub 2007 Sep 25. PMID 17895475
- [Background] van Rossum LG, van Rijn AF, Laheij RJ, van Oijen MG, Fockens P, van Krieken HH, Verbeek AL, Jansen JB, Dekker E. Random comparison of guaiac and immunochemical fecal occult blood tests for colorectal cancer in a screening population. Gastroenterology. 2008 Jul;135(1):82-90. doi: 10.1053/j.gastro.2008.03.040. Epub 2008 Mar 25. PMID 18482589
- [Background] Zorzi M, Fedeli U, Schievano E, Bovo E, Guzzinati S, Baracco S, Fedato C, Saugo M, Dei Tos AP. Impact on colorectal cancer mortality of screening programmes based on the faecal immunochemical test. Gut. 2015 May;64(5):784-90. doi: 10.1136/gutjnl-2014-307508. Epub 2014 Sep 1. PMID 25179811
- [Background] Bevolkingsonderzoek Darmkanker Monitor 2017. Erasmus MC en NKI / AvL; 2017
- [Background] de Wijkerslooth TR, Stoop EM, Bossuyt PM, Meijer GA, van Ballegooijen M, van Roon AH, Stegeman I, Kraaijenhagen RA, Fockens P, van Leerdam ME, Dekker E, Kuipers EJ. Immunochemical fecal occult blood testing is equally sensitive for proximal and distal advanced neoplasia. Am J Gastroenterol. 2012 Oct;107(10):1570-8. doi: 10.1038/ajg.2012.249. Epub 2012 Jul 31. PMID 22850431
- [Background] Cubiella J, Castro I, Hernandez V, Gonzalez-Mao C, Rivera C, Iglesias F, Cid L, Soto S, de-Castro L, Vega P, Hermo JA, Macenlle R, Martinez A, Martinez-Ares D, Estevez P, Cid E, Herreros-Villanueva M, Portillo I, Bujanda L, Fernandez-Seara J; COLONPREV study investigators. Characteristics of adenomas detected by fecal immunochemical test in colorectal cancer screening. Cancer Epidemiol Biomarkers Prev. 2014 Sep;23(9):1884-92. doi: 10.1158/1055-9965.EPI-13-1346. Epub 2014 Jun 24. PMID 24962836
- [Background] Wong MC, Ching JY, Chan VC, Lam TY, Shum JP, Luk AK, Wong SS, Ng SC, Ng SS, Wu JC, Chan FK, Sung JJ. Diagnostic Accuracy of a Qualitative Fecal Immunochemical Test Varies With Location of Neoplasia But Not Number of Specimens. Clin Gastroenterol Hepatol. 2015 Aug;13(8):1472-9. doi: 10.1016/j.cgh.2015.02.021. Epub 2015 Feb 24. PMID 25724708
- [Background] Dekker N, van Rossum LG, Van Vugt-van Pinxteren M, van Stiphout SH, Hermens RP, van Zelst-Stams WA, van Oijen MG, Laheij RJ, Jansen JB, Hoogerbrugge N. Adding familial risk assessment to faecal occult blood test can increase the effectiveness of population-based colorectal cancer screening. Eur J Cancer. 2011 Jul;47(10):1571-7. doi: 10.1016/j.ejca.2011.01.022. Epub 2011 Feb 28. PMID 21367600
- [Background] Cha JM, Lee JI, Joo KR, Shin HP, Park JJ, Jeun JW, Lim JU. First-degree relatives of colorectal cancer patients are likely to show advanced colorectal neoplasia despite a negative fecal immunochemical test. Digestion. 2012;86(4):283-7. doi: 10.1159/000341738. Epub 2012 Oct 9. PMID 23051697
- [Background] de Jong AE, Vasen HF. The frequency of a positive family history for colorectal cancer: a population-based study in the Netherlands. Neth J Med. 2006 Nov;64(10):367-70. PMID 17122453
- [Background] Lynch HT, de la Chapelle A. Hereditary colorectal cancer. N Engl J Med. 2003 Mar 6;348(10):919-32. doi: 10.1056/NEJMra012242. No abstract available. PMID 12621137
- [Background] Worthley DL, Smith A, Bampton PA, Cole SR, Young GP. Many participants in fecal occult blood test population screening have a higher-than-average risk for colorectal cancer. Eur J Gastroenterol Hepatol. 2006 Oct;18(10):1079-83. doi: 10.1097/01.meg.0000231754.35340.fa. PMID 16957514
- [Background] Regula J, Rupinski M, Kraszewska E, Polkowski M, Pachlewski J, Orlowska J, Nowacki MP, Butruk E. Colonoscopy in colorectal-cancer screening for detection of advanced neoplasia. N Engl J Med. 2006 Nov 2;355(18):1863-72. doi: 10.1056/NEJMoa054967. PMID 17079760
- [Background] Chang LC, Wu MS, Tu CH, Lee YC, Shun CT, Chiu HM. Metabolic syndrome and smoking may justify earlier colorectal cancer screening in men. Gastrointest Endosc. 2014 Jun;79(6):961-9. doi: 10.1016/j.gie.2013.11.035. Epub 2014 Jan 25. PMID 24472766
- [Background] Betes M, Munoz-Navas MA, Duque JM, Angos R, Macias E, Subtil JC, Herraiz M, De La Riva S, Delgado-Rodriguez M, Martinez-Gonzalez MA. Use of colonoscopy as a primary screening test for colorectal cancer in average risk people. Am J Gastroenterol. 2003 Dec;98(12):2648-54. doi: 10.1111/j.1572-0241.2003.08771.x. PMID 14687811
- [Background] Nguyen SP, Bent S, Chen YH, Terdiman JP. Gender as a risk factor for advanced neoplasia and colorectal cancer: a systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2009 Jun;7(6):676-81.e1-3. doi: 10.1016/j.cgh.2009.01.008. PMID 19514116
- [Background] Stegeman I, de Wijkerslooth TR, Stoop EM, van Leerdam ME, Dekker E, van Ballegooijen M, Kuipers EJ, Fockens P, Kraaijenhagen RA, Bossuyt PM. Colorectal cancer risk factors in the detection of advanced adenoma and colorectal cancer. Cancer Epidemiol. 2013 Jun;37(3):278-83. doi: 10.1016/j.canep.2013.02.004. Epub 2013 Mar 9. PMID 23491770
- [Background] Yeoh KG, Ho KY, Chiu HM, Zhu F, Ching JY, Wu DC, Matsuda T, Byeon JS, Lee SK, Goh KL, Sollano J, Rerknimitr R, Leong R, Tsoi K, Lin JT, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. The Asia-Pacific Colorectal Screening score: a validated tool that stratifies risk for colorectal advanced neoplasia in asymptomatic Asian subjects. Gut. 2011 Sep;60(9):1236-41. doi: 10.1136/gut.2010.221168. Epub 2011 Mar 14. PMID 21402615
- [Background] Ma GK, Ladabaum U. Personalizing colorectal cancer screening: a systematic review of models to predict risk of colorectal neoplasia. Clin Gastroenterol Hepatol. 2014 Oct;12(10):1624-34.e1. doi: 10.1016/j.cgh.2014.01.042. Epub 2014 Feb 15. PMID 24534546
- [Background] Aniwan S, Rerknimitr R, Kongkam P, Wisedopas N, Ponuthai Y, Chaithongrat S, Kullavanijaya P. A combination of clinical risk stratification and fecal immunochemical test results to prioritize colonoscopy screening in asymptomatic participants. Gastrointest Endosc. 2015 Mar;81(3):719-27. doi: 10.1016/j.gie.2014.11.035. PMID 25708760
- [Background] Robertson DJ, Imperiale TF. Stool Testing for Colorectal Cancer Screening. Gastroenterology. 2015 Oct;149(5):1286-93. doi: 10.1053/j.gastro.2015.05.045. Epub 2015 May 30. PMID 26033632
- [Background] Stegeman I, de Wijkerslooth TR, Stoop EM, van Leerdam ME, Dekker E, van Ballegooijen M, Kuipers EJ, Fockens P, Kraaijenhagen RA, Bossuyt PM. Combining risk factors with faecal immunochemical test outcome for selecting CRC screenees for colonoscopy. Gut. 2014 Mar;63(3):466-71. doi: 10.1136/gutjnl-2013-305013. Epub 2013 Aug 20. PMID 23964098
- [Background] Altman DG, Bland JM. Statistics notes. Treatment allocation in controlled trials: why randomise? BMJ. 1999 May 1;318(7192):1209. doi: 10.1136/bmj.318.7192.1209. No abstract available. PMID 10221955
- [Background] Colkesen EB, Ferket BS, Tijssen JG, Kraaijenhagen RA, van Kalken CK, Peters RJ. Effects on cardiovascular disease risk of a web-based health risk assessment with tailored health advice: a follow-up study. Vasc Health Risk Manag. 2011;7:67-74. doi: 10.2147/VHRM.S16340. Epub 2011 Feb 9. PMID 21415919
- [Background] Umar A, Boland CR, Terdiman JP, Syngal S, de la Chapelle A, Ruschoff J, Fishel R, Lindor NM, Burgart LJ, Hamelin R, Hamilton SR, Hiatt RA, Jass J, Lindblom A, Lynch HT, Peltomaki P, Ramsey SD, Rodriguez-Bigas MA, Vasen HF, Hawk ET, Barrett JC, Freedman AN, Srivastava S. Revised Bethesda Guidelines for hereditary nonpolyposis colorectal cancer (Lynch syndrome) and microsatellite instability. J Natl Cancer Inst. 2004 Feb 18;96(4):261-8. doi: 10.1093/jnci/djh034. PMID 14970275
- [Background] Rex DK. Quality in colonoscopy: cecal intubation first, then what? Am J Gastroenterol. 2006 Apr;101(4):732-4. doi: 10.1111/j.1572-0241.2006.00483.x. PMID 16635220
- [Background] Protocol voor de toelating en auditing van coloscopiecentra en endoscopisten. Rijksinstituut voor Volksgezondheid en Milieu; 2018
- [Background] Landelijke Monitoring en Evaluatie Bevolkingsonderzoek Darmkanker. In: Milieu RvVe, ed.2019
- [Background] Schlemper RJ, Riddell RH, Kato Y, Borchard F, Cooper HS, Dawsey SM, Dixon MF, Fenoglio-Preiser CM, Flejou JF, Geboes K, Hattori T, Hirota T, Itabashi M, Iwafuchi M, Iwashita A, Kim YI, Kirchner T, Klimpfinger M, Koike M, Lauwers GY, Lewin KJ, Oberhuber G, Offner F, Price AB, Rubio CA, Shimizu M, Shimoda T, Sipponen P, Solcia E, Stolte M, Watanabe H, Yamabe H. The Vienna classification of gastrointestinal epithelial neoplasia. Gut. 2000 Aug;47(2):251-5. doi: 10.1136/gut.47.2.251. PMID 10896917
- [Background] Nederlandse Richtlijn Coloscopie Surveillance. Nederlandse Vereniging van Maag-, Darm- en Levertartsen; 2013
- [Derived] Kortlever TL, van der Vlugt M, Duijkers FAM, Masclee A, Kraaijenhagen R, Spaander MCW, Lansdorp-Vogelaar I, Bossuyt PM, Dekker E. Diagnostic yield of a risk model versus faecal immunochemical test only: a randomised controlled trial in a colorectal cancer screening programme. Br J Cancer. 2023 Sep;129(5):791-796. doi: 10.1038/s41416-023-02358-z. Epub 2023 Jul 19. PMID 37468570